CLINICAL TRIAL: NCT00362232
Title: RECORD 4 Study: REgulation of Coagulation in ORthopedic Surgery to Prevent DVT and PE; a Controlled, Double-blind, Randomized Study of BAY59-7939 in the Prevention of VTE in Subjects Undergoing Elective Total Knee Replacement
Brief Title: Regulation of Coagulation in Orthopedic Surgery to Prevent Deep Vein Thromboembolism (DVT) and Pulmonary Embolism (PE). A Study of BAY59-7939 in the Prevention of Venous Thrombo Embolism (VTE) in Subjects Undergoing Elective Total Knee Replacement.
Acronym: RECORD 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11355; 2006-002402-60 (EudraCT Number)
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Results first posted 2012-06-13 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Venous Thromboembolism
Keywords: Prevention of venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban 10 mg Once Daily (OD) ((Xarelto, BAY59-7939)) (Experimental): Rivaroxaban (Xarelto, BAY59-7939) 10 mg tablet administered once daily (od) in the evening plus placebo syringes of enoxaparin twice a day (bid) administered once in the morning and once in the evening.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Placebo: syringes of Enoxaparin
- Enoxaparin 30 mg twice a day (bid) (Active Comparator): Placebo tablet of rivaroxaban administered once daily in the evening plus syringes of enoxaparin active substance 30 mg twice a day administered once in the morning and once in the evening.
  Interventions: Drug: Enoxaparin; Drug: Placebo: tablet of Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Rivaroxaban (Xarelto, BAY59-7939) 10 mg tablet administered once daily (od) in the evening.
  Arms: Rivaroxaban 10 mg Once Daily (OD) ((Xarelto, BAY59-7939))
Drug: Enoxaparin — Syringes of enoxaparin active substance 30 mg twice a day administered once in the morning and once in the evening.
  Arms: Enoxaparin 30 mg twice a day (bid)
Drug: Placebo: tablet of Rivaroxaban — Placebo tablet of rivaroxaban administered once daily in the evening.
  Arms: Enoxaparin 30 mg twice a day (bid)
Drug: Placebo: syringes of Enoxaparin — Placebo syringes of enoxaparin twice a day (bid) administered once in the morning and once in the evening.
  Arms: Rivaroxaban 10 mg Once Daily (OD) ((Xarelto, BAY59-7939))

SUMMARY:
The purpose of this study is to assess if 10 mg BAY59-7939, taken once daily as a tablet, is safe and prevents blood clot which may form after a knee replacement operation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years or above
* Patients scheduled for elective total knee replacement

Exclusion Criteria:

* Active bleeding or high risk of bleeding contraindicating treatment with Low Molecular Weight Heparin (LMWH)
* Contraindication listed in the labeling or conditions precluding subject treatment with enoxaparin or requiring dose adjustment (e.g. severe renal impairment, please refer to the local label of enoxaparin in your country)
* Conditions prohibiting bilateral venography (e.g. amputation of 1 leg, allergy to contrast media)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3148 (Actual)
Dates: Start 2006-06; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (113):
- United States (39):
  - Birmingham, Alabama
  - Tuscaloosa, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Bakersfield, California
  - Encinitas, California
  - Fountain Valley, California
  - La Jolla, California
  - Torrance, California
  - Yuba City, California
  - Centennial, Colorado
  - Denver, Colorado
  - Englewood, Colorado
  - Boynton Beach, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Pensacola, Florida
  - Pinellas Park, Florida
  - Decatur, Georgia
  - Boise, Idaho
  - Meridian, Idaho
  - Towson, Maryland
  - Missoula, Montana
  - Teaneck, New Jersey
  - Greensboro, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Johnstown, Pennsylvania
  - State College, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Grapevine, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Spokane, Washington
- Bulgaria (3):
  - Pleven
  - Plovdiv
  - Sofia
- Canada (16):
  - Red Deer, Alberta
  - Kelowna, British Columbia
  - Penticton, British Columbia
  - Fredericton, New Brunswick
  - Ajax, Ontario
  - Brantford, Ontario
  - Greater Sudbury, Ontario
  - Oakville, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Peterborough, Ontario
  - Scarborough Village, Ontario
  - Thunder Bay, Ontario
  - Woodstock, Ontario
  - Charlottetown, Prince Edward Island
  - Montreal, Quebec
- Denmark (6):
  - Hellerup
  - Herlev
  - Hvidovre
  - Hørsholm
  - Silkeborg
  - Viborg
- India (11):
  - Hyderabad, Andhra Pradesh
  - Secunderabad, Andhra Pradesh
  - Secundrabad, Andhra Pradesh
  - Ahmedabad, Gujarat
  - Pune, Maharashtra
  - Ludhiana, Punjab
  - Chennai, Tamil Nadu
  - Bangalore
  - Baroda
  - Hyderabad
  - New Delhi
- Israel (6):
  - Petah Tikva, Israel
  - Ẕerifin, Israel
  - Beersheba
  - Holon
  - Kfar Saba
  - Tel Aviv
- Lithuania (4):
  - Kaunas
  - Klaipėda
  - Panevezys
  - Vilnius
- Mexico (5):
  - Guadalajara, Jalisco
  - Zapopan, Jalisco
  - Monterrey, Nuevo León
  - Mérida, Yucatán
  - Edo. de Mexico
- Norway (4):
  - Baerum Postterminal
  - Gjøvik
  - Kongsvinger
  - Lillehammer
- Karachi, Sindh, Pakistan
- Poland (9):
  - Bydgoszcz
  - Elblag
  - Gdansk
  - Gmina Końskie
  - Kielce
  - Krakow
  - Lublin
  - Sosnowiec
  - Warsaw
- Sri Lanka (3):
  - Colombo-80
  - Ragama
  - Sri Jayewardenepura Kotte
- Sweden (6):
  - Gothenburg
  - Hässleholm
  - Örebro
  - Stockholm
  - Vaxjo
  - Västervik

REFERENCES:
- [Result] Turpie AG, Lassen MR, Davidson BL, Bauer KA, Gent M, Kwong LM, Cushner FD, Lotke PA, Berkowitz SD, Bandel TJ, Benson A, Misselwitz F, Fisher WD; RECORD4 Investigators. Rivaroxaban versus enoxaparin for thromboprophylaxis after total knee arthroplasty (RECORD4): a randomised trial. Lancet. 2009 May 16;373(9676):1673-80. doi: 10.1016/S0140-6736(09)60734-0. Epub 2009 May 4. PMID 19411100
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from 16 Jun 2006 to 31 Jan 2008.
Pre-assignment Details: 3418 subjects were screened; 270 subjects were screening failures and were not randomized; 3148 subjects were randomized; 114 subjects did not receive medication; 3034 subjects received medication and were included in the safety population
Groups:
- Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939): Rivaroxaban (Xarelto, BAY59-7939) 10 mg tablet administered once daily (od) in the evening plus placebo syringes of enoxaparin twice a day (bid) administered once in the morning and once in the evening.
Period: Treatment (12 +/- 2 Days)
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Started | 1584 | 1564
Received Treatment | 1526 (Safety population) | 1508 (Safety population)
Completed | 1425 | 1413
Not Completed | 159 | 151
Not completed — Adverse Event | 62 | 56
Not completed — Death | 1 | 3
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 2 | 5
Not completed — Protocol Violation | 22 | 21
Not completed — Withdrawal by Subject | 49 | 47
Not completed — Noncompliance to Study Drug | 9 | 0
Not completed — Technical Problems | 1 | 0
Not completed — Clinical Endpoint Reached | 10 | 18
Period: Follow-up (30 (+ 5) Days)
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Started | 1471 | 1455
Completed | 1433 | 1416
Not Completed | 38 | 39
Not completed — Adverse Event | 2 | 3
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 27 | 28
Not completed — Withdrawal by Subject | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid) | Total
Number analyzed (Participants) | 1526 | 1508 | 3034
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (9.7) | 64.7 (9.7) | 64.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1007 | 967 | 1974
  Male | 519 | 541 | 1060
Race/Ethnicity, Customized [Number; unit: participants] — One subject in the rivaroxaban 10 mg OD treatment group was missing race.
  participants
    White | 1008 | 1032 | 2040
    Black | 88 | 65 | 153
    Asian | 289 | 289 | 578
    American Indian | 1 | 4 | 5
    Hispanic | 137 | 116 | 253
    Uncodable | 2 | 2 | 4
Weight [Number; unit: participants] — One subject in each treatment group was missing baseline weight.
  participants
    =< 50 kg | 22 | 28 | 50
    > 50 - 70 kg | 367 | 358 | 725
    > 70 - 90 kg | 629 | 616 | 1245
    > 90 - 110 kg | 322 | 343 | 665
    > 110 kg | 185 | 162 | 347

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint of Total Venous Thrombo Embolism (VTE) i.e.: Any Deep Vein Thromboembolism (DVT) (Proximal and/or Distal), Non Fatal Pulmonary Embolism (PE), Death of All Causes Per Protocol Population
Description: Blinded, adjudicated assessment of bilateral venography, clinical signs of deep vein thrombosis (DVT) and pulmonary embolism (PE), ultrasound, clinical chemistry and coagulation factors, autopsy report, electrocardiogram (ECG), pulmonary angiography, perfusion/ventilation lung scintigraphy, chest radiography, computed tomography
Time Frame: Up to 16 days after surgery
Population: The primary efficacy analysis was based on the per protocol (PP) population and included subjects who were valid for the modified intent to treat (MITT) population, had an adequate assessment of thromboembolism that, in case of a positive finding, was done not later than 36 hours after stop of study drug, and had no major protocol deviations.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 864 | 878
Percentage of participants | 6.71 | 9.34
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Null hypothesis: rivaroxaban is inferior to the comparator, ie, the incidence of the primary efficacy endpoint in the rivaroxaban group is larger by more than 4% (absolute) compared to the comparator group; Test type: Non-Inferiority or Equivalence — P-values were calculated based on the Mantel-Haenszel weighted estimator (one-sided); p < 0.001, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -2.71, 95% CI [-5.25 to -0.17] — Mantel-Haenszel weighted difference to Enoxaparin
Statistical Analysis 2: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Null hypothesis: The incidence of the primary efficacy endpoint is equal in the rivaroxaban group and the comparator group. P-values were calculated based on the Mantel-Haenszel weighted estimator (two-sided); Test type: Superiority or Other; p = 0.036, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -2.71, 95% CI [-5.25 to -0.17]

2. Primary Outcome: Composite Endpoint of Total VTE i.e.: Any DVT (Proximal and/or Distal), Non Fatal PE, Death of All Causes Per Modified Intent to Treat Population.
Description: as for outcome 1
Time Frame: Up to 16 days after surgery
Population: A subject was considered valid for the MITT analysis if the subject was valid for the safety analysis, had undergone the appropriate surgery, and had an adequate assessment of thromboembolism
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 965 | 959
Percentage of participants | 6.94 | 10.11
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.012, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -3.19, 95% CI [-5.67 to -0.71] — Mantel-Haenszel weighted difference to Enoxaparin

3. Secondary Outcome: Incidence of the Composite Endpoint Comprising Proximal DVT, Non-fatal PE and VTE- Related Death (Major VTE) Per Protocol Population of Major VTE
Description: as for outcome 1
Time Frame: Up to 16 days after surgery
Population: The PP population included subjects who were valid for the modified intent to treat (MITT) population, had an adequate assessment of thromboembolism that, in case of a positive finding, was done not later than 36 hours after stop of study drug, and had no major protocol deviations.
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 1011 | 1020
percentage of participants | 1.09 | 1.47
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Null hypothesis: The incidence of the major VTE is equal in the rivaroxaban group and the comparator group. P-values were calculated based on the Mantel-Haenszel weighted estimator (two-sided); Test type: Superiority or Other; p = 0.456, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -0.37, 95% CI [-1.34 to 0.6] — Mantel-Haenszel weighted difference to Enoxaparin
Statistical Analysis 2: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Null hypothesis: rivaroxaban is inferior to the comparator, ie, the incidence of the major VTE in the rivaroxaban group is larger by more than 1.5% (absolute) compared to the comparator group; Test type: Non-Inferiority or Equivalence — P-values were calculated based on the Mantel-Haenszel weighted estimator (one-sided); p < 0.001, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -0.37, 95% CI [-1.34 to 0.6]

4. Secondary Outcome: Incidence of the Composite Endpoint Comprising Proximal DVT, Non-fatal PE and VTE- Related Death (Major VTE) Per Modified Intent to Treat Population of Major VTE.
Description: as for outcome 1
Time Frame: Up to 16 days after surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 1122 | 1112
percentage of participants | 1.16 | 1.98
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.124, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -0.80, 95% CI [-1.82 to 0.22] — Mantel-Haenszel weighted difference to Enoxaparin
Statistical Analysis 2: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); [analysis description as in outcome 3, analysis 2]; Test type: Non-Inferiority or Equivalence — P-values were calculated based on the Mantel-Haenszel weighted estimator (one-sided); p < 0.001, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -0.80, 95% CI [-1.82 to 0.22]

5. Secondary Outcome: Incidence of Symptomatic VTE (DVT, PE) Per Protocol Population.
Description: Blinded, adjudicated assessment of bilateral venography, clinical signs of DVT and PE, ultrasound, clinical chemistry and coagulation factors, autopsy report, electrocardiogram (ECG), pulmonary angiography, perfusion/ventilation lung scintigraphy, chest radiography, computed tomography
Time Frame: Up to 16 days after surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 864 | 878
percentage of participants | 1.04 | 1.48
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Test type: Superiority or Other; Risk Difference (RD) = -0.44, 95% CI [-1.59 to 0.66] — Mantel-Haenszel weighted difference to Enoxaparin

6. Secondary Outcome: Incidence of Symptomatic VTE (DVT, PE) Per Modified Intent to Treat Population.
Description: as for outcome 5
Time Frame: Up to 16 days after surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 965 | 959
percentage of participants | 1.14 | 1.88
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Test type: Superiority or Other; Risk Difference (RD) = -0.72, 95% CI [-1.81 to 0.36] — Mantel-Haenszel weighted difference to Enoxaparin

7. Secondary Outcome: Incidence of DVT (Proximal, Distal) Per Protocol Population.
Description: as for outcome 5
Time Frame: Up to 16 days after surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 864 | 878
percentage of participants | 6.37 | 8.66
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Test type: Superiority or Other; Risk Difference (RD) = -2.38, 95% CI [-4.84 to 0.07] — Mantel-Haenszel weighted difference to Enoxaparin

8. Secondary Outcome: Incidence of DVT (Proximal, Distal) Per Modified Intent to Treat Population.
Description: as for outcome 5
Time Frame: Up to 16 days after surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 965 | 959
percentage of participants | 6.32 | 8.97
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Test type: Superiority or Other; Risk Difference (RD) = -2.67, 95% CI [-5.02 to -0.32] — Mantel-Haenszel weighted difference to Enoxaparin

9. Secondary Outcome: Incidence of Symptomatic VTE During Follow-up Per Protocol Population.
Description: as for outcome 5
Time Frame: Up to 47 days after surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 864 | 878
percentage of participants | 0.35 | 0.11
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Test type: Superiority or Other; Risk Difference (RD) = 0.24, 95% CI [-0.22 to 0.71] — Mantel-Haenszel weighted difference to Enoxaparin

10. Secondary Outcome: Incidence of Symptomatic VTE During Follow-up Per Modified Intent to Treat Population.
Description: as for outcome 5
Time Frame: Up to 47 days after surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 965 | 959
percentage of participants | 0.31 | 0.21
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Test type: Superiority or Other; Risk Difference (RD) = 0.11, 95% CI [-0.35 to 0.56]

11. Secondary Outcome: The Composite Endpoint Comprising Major VTE and Treatment-emergent Major Bleeding Per Subjects Valid for Analysis of Net Clinical Benefit
Description: Blinded, adjudicated assessment of bilateral venography, clinical signs of DVT and PE, ultrasound, clinical chemistry and coagulation factors, autopsy report, electrocardiogram (ECG), pulmonary angiography, perfusion/ventilation lung scintigraphy, chest radiography, computed tomography, anesthesia and surgery reports, number of transfusions
Time Frame: Up to 47 days after surgery
Population: The net clinical benefit population comprised all subjects either valid for MITT analysis of major VTE or who showed treatment-emergent major bleeding.
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 1130 | 1114
percentage of participants | 2.04 | 2.33
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Test type: Superiority or Other; Risk Difference (RD) = -0.30, 95% CI [-1.56 to 0.94] — Exact methods for difference to Enoxaparin

12. Secondary Outcome: Incidence of the Composite Endpoint That Results From the Primary Endpoint by Substituting VTE Related Death for All Death Per Protocol Population.
Description: as for outcome 5
Time Frame: Up to 16 days after surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 864 | 878
percentage of participants | 6.71 | 9.11
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Null hypothesis: The incidence rate is equal in the rivaroxaban group and the comparator group. P-values were calculated based on the Mantel-Haenszel weighted estimator (two-sided); Test type: Superiority or Other; p = 0.054, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -2.47, 95% CI [-4.99 to 0.04] — Mantel-Haenszel weighted difference to Enoxaparin
Statistical Analysis 2: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Null hypothesis: rivaroxaban is inferior to the comparator, ie, the incidence rate in the rivaroxaban group is larger by more than 4% (absolute) compared to the comparator group; Test type: Non-Inferiority or Equivalence — P-values were calculated based on the Mantel-Haenszel weighted estimator (one-sided); p < 0.001, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -2.47, 95% CI [-4.49 to 0.04]

13. Secondary Outcome: Incidence of the Composite Endpoint That Results From the Primary Endpoint by Substituting VTE Related Death for All Death Per Modified Intent to Treat Population.
Description: as for outcome 5
Time Frame: Up to 16 days after surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 965 | 959
percentage of participants | 6.84 | 9.80
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.017, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -2.97, 95% CI [-5.42 to -0.53] — Mantel-Haenszel weighted difference to Enoxaparin
Statistical Analysis 2: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); [analysis description as in outcome 12, analysis 2]; Test type: Non-Inferiority or Equivalence — P-values were calculated based on the Mantel-Haenszel weighted estimator (one-sided); p < 0.001, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -2.97, 95% CI [-5.42 to -0.53]

14. Secondary Outcome: Incidence of the Composite Endpoint That Results From Major VTE by Substituting All Cause Mortality for VTE-related Death Per Protocol of Major VTE Population.
Description: as for outcome 5
Time Frame: Up to 16 days after surgery
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 1011 | 1020
percentage of participants | 1.09 | 1.67
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.270, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -0.57, 95% CI [-1.57 to 0.44] — Mantel-Haenszel weighted difference to Enoxaparin
Statistical Analysis 2: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); Null hypothesis: rivaroxaban is inferior to the comparator, ie, the incidence rate in the rivaroxaban group is larger by more than 1.5% (absolute) compared to the comparator group; Test type: Non-Inferiority or Equivalence — P-values were calculated based on the Mantel-Haenszel weighted estimator (one-sided); p < 0.001, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -0.57, 95% CI [-1.57 to 0.44]

15. Secondary Outcome: Incidence of the Composite Endpoint That Results From Major VTE by Substituting All Cause Mortality for VTE-related Death Per Modified Intent to Treat of Major VTE Population.
Description: as for outcome 5
Time Frame: Up to 16 days after surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 1122 | 1112
percentage of participants | 1.25 | 2.25
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.074, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -0.98, 95% CI [-2.06 to 0.10] — Mantel-Haenszel weighted difference to Enoxaparin
Statistical Analysis 2: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); [analysis description as in outcome 14, analysis 2]; Test type: Non-Inferiority or Equivalence — P-values were calculated based on the Mantel-Haenszel weighted estimator (one-sided); p < 0.001, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = -0.98, 95% CI [-2.06 to 0.10]

16. Secondary Outcome: Treatment-emergent Major Bleedings Per Safety Population.
Description: Blinded, adjudicated assessments of all available information (eg, anesthesia and surgery reports, laboratory results, number of transfusions, autopsy report)
Time Frame: from start of double-blind study medication to last dose of double-blind study medication plus two days. The average duration of double-blind treatment was 12 days in each treatment group (safety population).
Population: The safety population comprised those subjects who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Number analyzed (Participants) | 1526 | 1508
percentage of participants | 0.66 | 0.27
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) vs Enoxaparin 30 mg Twice a Day (Bid); [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.110, Mantel Haenszel; weighted treatment differences; Risk Difference (RD) = 0.39, 95% CI [-0.09 to 0.88] — Mantel-Haenszel weighted difference to Enoxaparin

ADVERSE EVENTS:
Arm/Group | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) | Enoxaparin 30 mg Twice a Day (Bid)
Serious Adverse Events (participants affected / at risk) | 106/1526 | 131/1508
Other Adverse Events (participants affected / at risk) | 1167/1526 | 1152/1508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) (N=1526) | Enoxaparin 30 mg Twice a Day (Bid) (N=1508)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocythaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 4
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 6
Adrenal haemorrhage (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 3
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3
Chest pain (General disorders) | 3 | 6
Death (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 4
Pyrexia (General disorders) | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 3 | 9
Cellulitis (Infections and infestations) | 4 | 4
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 3 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 6
Post procedural infection (Infections and infestations) | 0 | 3
Postoperative wound infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 3 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Wound infection (Infections and infestations) | 2 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Device malfunction (Injury, poisoning and procedural complications) | 0 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 2 | 3
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 1
Clostridium difficile toxin test positive (Investigations) | 1 | 0
Coagulation factor increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 2
International normalised ratio increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 2 | 0
Occult blood positive (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fluctuance (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 2
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Peroneal nerve palsy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 2 | 0
Delirium tremens (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 5 | 4
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Urethral caruncle (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 13 | 22
Embolism venous (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 3 | 3
Haemorrhage (Vascular disorders) | 3 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Wound haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban 10 mg Once Daily (OD) (Xarelto, BAY59-7939) (N=1526) | Enoxaparin 30 mg Twice a Day (Bid) (N=1508)
Anaemia (Blood and lymphatic system disorders) | 57 | 51
Thrombocythaemia (Blood and lymphatic system disorders) | 33 | 35
Bradycardia (Cardiac disorders) | 15 | 16
Tachycardia (Cardiac disorders) | 96 | 95
Abdominal pain (Gastrointestinal disorders) | 21 | 13
Abdominal pain upper (Gastrointestinal disorders) | 16 | 16
Constipation (Gastrointestinal disorders) | 258 | 266
Diarrhoea (Gastrointestinal disorders) | 61 | 55
Dyspepsia (Gastrointestinal disorders) | 42 | 46
Hyperchlorhydria (Gastrointestinal disorders) | 9 | 17
Nausea (Gastrointestinal disorders) | 272 | 282
Vomiting (Gastrointestinal disorders) | 157 | 131
Asthenia (General disorders) | 77 | 84
Chest pain (General disorders) | 16 | 24
Chills (General disorders) | 28 | 33
Fatigue (General disorders) | 79 | 79
Oedema (General disorders) | 43 | 38
Oedema peripheral (General disorders) | 235 | 256
Pain (General disorders) | 19 | 25
Pyrexia (General disorders) | 320 | 310
Urinary tract infection (Infections and infestations) | 40 | 39
Anaemia postoperative (Injury, poisoning and procedural complications) | 178 | 187
Contusion (Injury, poisoning and procedural complications) | 27 | 31
Post procedural swelling (Injury, poisoning and procedural complications) | 16 | 11
Procedural nausea (Injury, poisoning and procedural complications) | 26 | 22
Procedural pain (Injury, poisoning and procedural complications) | 172 | 186
Wound secretion (Injury, poisoning and procedural complications) | 19 | 15
Alanine aminotransferase increased (Investigations) | 24 | 45
Aspartate aminotransferase increased (Investigations) | 22 | 28
Blood alkaline phosphatase increased (Investigations) | 14 | 21
Blood creatinine increased (Investigations) | 17 | 18
Blood lactate dehydrogenase increased (Investigations) | 33 | 29
Blood potassium decreased (Investigations) | 19 | 24
Body temperature increased (Investigations) | 63 | 81
Breath sounds abnormal (Investigations) | 22 | 22
Gamma-glutamyltransferase increased (Investigations) | 40 | 52
Haemoglobin decreased (Investigations) | 44 | 33
Lipase increased (Investigations) | 16 | 17
Anorexia (Metabolism and nutrition disorders) | 18 | 28
Decreased appetite (Metabolism and nutrition disorders) | 16 | 19
Hypokalaemia (Metabolism and nutrition disorders) | 41 | 53
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 | 67
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 21
Joint swelling (Musculoskeletal and connective tissue disorders) | 35 | 39
Joint warmth (Musculoskeletal and connective tissue disorders) | 21 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 96 | 88
Pain in extremity (Musculoskeletal and connective tissue disorders) | 131 | 119
Dizziness (Nervous system disorders) | 111 | 102
Headache (Nervous system disorders) | 49 | 46
Hypoaesthesia (Nervous system disorders) | 30 | 38
Lethargy (Nervous system disorders) | 16 | 13
Somnolence (Nervous system disorders) | 64 | 58
Anxiety (Psychiatric disorders) | 44 | 39
Confusional state (Psychiatric disorders) | 38 | 35
Insomnia (Psychiatric disorders) | 163 | 168
Dysuria (Renal and urinary disorders) | 19 | 12
Pollakiuria (Renal and urinary disorders) | 20 | 11
Urinary retention (Renal and urinary disorders) | 72 | 65
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 39
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47 | 36
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 | 19
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 26 | 26
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 | 26
Wheezing (Respiratory, thoracic and mediastinal disorders) | 15 | 21
Blister (Skin and subcutaneous tissue disorders) | 37 | 25
Ecchymosis (Skin and subcutaneous tissue disorders) | 28 | 31
Erythema (Skin and subcutaneous tissue disorders) | 79 | 75
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 18 | 24
Pruritus (Skin and subcutaneous tissue disorders) | 128 | 123
Pruritus generalised (Skin and subcutaneous tissue disorders) | 20 | 14
Rash (Skin and subcutaneous tissue disorders) | 36 | 40
Deep vein thrombosis (Vascular disorders) | 52 | 68
Hypertension (Vascular disorders) | 34 | 21
Hypotension (Vascular disorders) | 100 | 102
Thrombosis (Vascular disorders) | 25 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No